CLINICAL TRIAL: NCT05912335
Title: Clinical Efficiency of Xanthan Hydrogels Containing Local Anesthetics Encapsulated in Nanostructured Lipid Carries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Michelle Franz Montan Braga Leite, DDS, MSc, PhD, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CAAE: 45317521.9.0000.5418
Record Dates: First submitted 2023-05-25; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Dental Trauma; Local Anesthesia; Oral Cavity Disease
Keywords: Topical Anesthesia; Topical Formulation; Oral Mucosa; Lidocaine; Prilocaine; Nanostructured Lipid Carrier
MeSH Terms: conditions — Mouth Diseases | interventions — Anesthetics, Local; Dosage Forms

STUDY DESIGN:
Intervention Model Description: 40 volunteers will receive the following formulations: hydrogels containing LAs - lidocaine, and prilocaine (both at 2.5%) encapsulated in CLN (XAN-CLN) or not (XAN-CLN ), EMLA and placebo hydrogel. The formulations will be applied for 2 minutes, bilaterally on the palatal mucosa (first premolar region), in two distinct sessions. Soon after the removal of the topical formulation, an AL will be performed at the region using 0.3 mL of anesthetic solution at an injection speed of 1 mL/min. Pain resulting from needle insertion and LA injection will be measured using two visual analog scales (VAS).
Who Masked: Participant, Care Provider
Masking Description: The participant and the applicator don't know which formulation was applied because these were named A, B, C, and D and the applicator doesn't have access to the data of which formulation was titled by each letter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Topical anesthetic available on the market - Lidocaine (2.5%), Prilocaine (2.5%) (Active Comparator): Applied at palatal mucosa (first premolar region), for 2 minutes. After that, this formulation will be removed.
  100 mg.
  Interventions: Drug: Topical anesthetic
- Xanthan hydrogel 2% (Placebo Comparator): Applied at palatal mucosa (first premolar region), for 2 minutes. After that, this formulation will be removed.
  100 mg.
  Interventions: Drug: Topical anesthetic
- Xanthan hydrogel (2%), Lidocaine (2.5%), Prilocaine (2.5%) in NLC (Experimental): Applied at palatal mucosa (first premolar region), for 2 minutes. After that, this formulation will be removed.
  100 mg. Local Anesthetic encapsulated in nanostructured lipid carriers (NLC)
  Interventions: Drug: Topical anesthetic
- Xanthan hydrogel (2%), Lidocaine (2.5%), Prilocaine (2.5%) (Experimental): Applied at palatal mucosa (first premolar region), for 2 minutes. After that, this formulation will be removed.
  100 mg.
  Interventions: Drug: Topical anesthetic

INTERVENTIONS:
Drug: Topical anesthetic — The topical anesthetic, or topical formulation, was applied to the palatal mucosa for 2 minutes.
  Other Names: Topical Formulation

SUMMARY:
In a crossover, randomized, placebo-controlled, double-blind study, 40 volunteers will receive the following formulations: hydrogels containing LAs (local anesthetic) - lidocaine and prilocaine (both at 2.5%) encapsulated in CLN (XAN-CLN) or not (XAN-CLN ), EMLA (topical anesthetic available on the market) and placebo hydrogel. The formulations will be applied for 2 minutes, bilaterally on the palatal mucosa (first premolar region), in two distinct sessions. Soon after removal of the topical formulation, an AL will be performed at the region using 0.3 mL of anesthetic solution at an injection speed of 1 mL/min. Pain resulting from needle insertion and LA injection will be measured using two visual analog scales (VAS).

DETAILED DESCRIPTION:
Dental treatment presents numerous innovations, but the pain associated with the administration of local anesthesia (LA) continuous to be a traumatic procedure for many patients. Although we use topical anesthetics (TA) to reduce pain, the commercially available formulations are only effective in preventing the pain of the needle puncture.

This project aims to evaluate the clinical efficacy of xanthan-based hydrogels (2%) containing LAs encapsulated in nanostructured lipid carriers (CLN), reducing pain during puncture and injection of LA in the palatine mucosa. In a crossover, randomized, placebo-controlled, double-blind study, 40 volunteers will receive the following formulations: hydrogels containing LAs - lidocaine and prilocaine (both at 2.5%) encapsulated in CLN (XAN-CLN) or not (XAN-CLN ), EMLA and placebo hydrogel. The formulations will be applied for 2 minutes, bilaterally on the palatal mucosa (first premolar region), in two distinct sessions. Soon after the removal of the topical formulation, an AL will be performed at the region using 0.3 mL of anesthetic solution at an injection speed of 1 mL/min. The computerized Morpheus® anesthetic injector will be used in order to control the variables of volume and injection speed. Pain resulting from needle insertion and LA injection will be measured using two visual analog scales (VAS). Hydrogels containing CLN are expected to have good mechanical properties and allow the permeation of LAs efficiently through the oral mucosal epithelium. In addition, they can improve the efficacy of topical anesthesia in order to perform a painless LA in the palatal mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* No lesions in the study area
* Have already been submitted to local anesthesia without intercurrence

Exclusion Criteria:

* Used any drugs that change the pain sensibility 1 week before
* Smokers
* Alcoholic

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Pain sensitivity assessment by Visual Analogue Scale after the puncture of the needle of the local anesthetic. | 2 minutes
  The blind investigator evaluated the values obtained on VAS, with a rule, the left far end mean 0, for no pain at all and the right far end mean 100 for maximum pain. Therefore, a a higher score means a worse outcome.

SECONDARY OUTCOMES:
Pain sensitivity assessment by Visual Analogue Scale after the injection of the local anesthetic. | 2 minutes
  The blind investigator evaluated the values obtained on VAS, with a rule, the left far end mean 0, for no pain at all and the right far end mean 100 for maximum pain. Therefore, a a higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Michelle Franz Montan Braga Leite, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No